CLINICAL TRIAL: NCT07393737
Title: The Effect of Virtual Reality Goggles and the Kaleidoscope Application During Renal Scintigraphy on Children's Fear and Anxiety Levels
Brief Title: The Effect of Using Virtual Reality and Kaleidoscope During Renal Scintigraphy on Children's Fear and Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Hüsniye ÇEKİÇ, Associate Professor, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5C679852b7f3
Record Dates: First submitted 2025-12-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Fear Anxiety
Keywords: fear anxiety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no intervention routine application group (No Intervention): No distraction techniques were used with the children in this group. They were informed about the routine imaging procedure at the clinic and their parents were allowed to stay with them during the imaging.
- kaleidoscope group (Experimental): During the scintigraphy scan (maximum 10 minutes), the children in this group had their attention diverted elsewhere using a kaleidoscope.
  Interventions: Other: kaleidoscope
- virtual reality group (Experimental): Children in this group were shown a cartoon featuring animals using virtual reality goggles. The video was started as soon as the child was placed on the scintigraphy device and continued until the scan was complete. The virtual reality goggles were removed once the scan was finished. Since the scan lasted a maximum of 10 minutes, care was taken to ensure that the selected video was at least 10 minutes long. Children who were given VR goggles were shown the cartoon "Smart Rabbit Momo." This process took an average of 10-15 minutes.
  Interventions: Other: virtual reality glasses

INTERVENTIONS:
Other: kaleidoscope — for use in nuclear medicine
  Arms: kaleidoscope group
Other: virtual reality glasses — The use of virtual reality in nuclear medicine
  Arms: virtual reality group

SUMMARY:
The kidneys are two bean-shaped organs that play a very important role in the human body. They are located on the right and left sides of the body, in the lower back. Their main function is to filter excess water and waste from the blood and excrete it through urine. Thus, they help maintain the body's fluid and electrolyte balance. They produce hormones that regulate blood pressure. They secrete the hormone erythropoietin, which stimulates the production of red blood cells. They play an important role in vitamin D metabolism to support bone health. Kidney scintigraphy is an important imaging method used to assess the function and structure of the kidneys. Using a radioactive substance, this test helps to examine the kidneys' blood flow, filtration and urine production. It is used to see how healthy the kidneys are working. It can help identify problems such as a mass or infection in the kidneys. It is used to detect urinary tract blockages caused by stones, tumors or other causes. It is important in patients who have had a kidney transplant to check that the new kidney is working properly. DMSA scintigraphy (Dimercaptosuccinic Acid scintigraphy) is a nuclear medicine imaging method used to assess the function and structural integrity of the kidneys. During imaging, the patient must remain immobile for a certain period of time, which can be difficult for children. Developing effective methods to divert children's attention and facilitate their adaptation to the hospital environment is of great importance in reducing both the comfort of patients and the workload of healthcare professionals. Virtual reality (VR) goggles are a highly effective tool for distraction. Because it engages our senses so intensely, it can cause us to largely ignore what is happening in the environment. VR goggles are very good at minimizing distractions or immersing you in a completely different atmosphere. The kaleidoscope is an impressive tool for diverting attention. Thanks to its mirrors and colored parts, it creates ever-changing and fascinating patterns. The hypnotic effect of the visual flow can relax the mind and help distract attention from stressful elements.

ELIGIBILITY:
Inclusion Criteria: Being between 4 and 6 years of age

* Speaking Turkish
* Having no communication problems
* Administration of radiopharmaceutical medication to the child prior to imaging
* Voluntary participation of the child and parent in the study

Exclusion Criteria: Not being between 4-6 years of age

* Having a chronic disease other than a kidney abnormality
* Having previously undergone a kidney scintigraphy scan
* One of the parents having previously undergone a kidney scintigraphy scan
* The child having a visual, hearing, or mental disability

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-08 (Estimated)

PRIMARY OUTCOMES:
The effect of virtual reality glasses and kaleidoscope application on children's fear and anxiety levels during renal scintigraphy. | about six months

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus Üniversitesi, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No